CLINICAL TRIAL: NCT06713252
Title: Art Therapy and Its Effect on Non-Motor Function Rehabilitation in the Subacute Phase of Stroke Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University (Other)
Responsible Party: Principal Investigator, Zexi Liu, Director, Chonbuk National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-23-24-048934
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Art Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art therapy (Experimental): Through music, painting, dance and other forms, art therapy can not only help patients regulate their emotions, relieve anxiety and depression, but also activate different areas of the brain to promote neuroplasticity, thereby promoting the recovery of motor function
  Interventions: Behavioral: Art therapy
- Regular therapy (Active Comparator): Standard treatment
  Interventions: Behavioral: Regular therapy

INTERVENTIONS:
Behavioral: Art therapy — Through music, painting, dance and other forms, art therapy can not only help patients regulate their emotions, relieve anxiety and depression, but also activate different areas of the brain to promote neuroplasticity, thereby promoting the recovery of motor function
  Arms: Art therapy
Behavioral: Regular therapy — Standard treatment
  Arms: Regular therapy

SUMMARY:
Stroke is one of the leading causes of disability and death worldwide, with the number of stroke patients steadily increasing due to the aging population. While traditional rehabilitation methods, such as pharmacological treatment, physical therapy, and cognitive therapy, can improve physical function to some extent, many stroke patients still face long-term non-motor impairments, including deficits in emotional, cognitive, and social functioning. Art therapy, as an integrative, non-invasive intervention, has gradually gained attention from researchers and clinicians due to its potential for restoring non-motor functions. Through artistic modalities such as music, painting, and dance, art therapy not only helps patients regulate their emotions, reducing anxiety and depression, but also promotes neuroplasticity, improving cognitive function and social participation. In the rehabilitation of stroke patients in the subacute phase, art therapy can serve as an adjunctive intervention, providing multidimensional rehabilitation support, optimizing emotional regulation and cognitive recovery, and offering new hope for the patients' overall rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Study Participants: Stroke patients aged 40-75. Patients in this age group generally have a higher incidence of stroke and show relatively higher plasticity during the rehabilitation process.
2. Type of Stroke: First occurrence of ischemic or hemorrhagic stroke, confirmed by imaging (CT or MRI). This helps to ensure consistency in the type of stroke among participants, reducing rehabilitation differences caused by varying stroke types.
3. Time Since Stroke Onset: Between 2 weeks and 3 months post-stroke (broadly defined subacute phase). During this phase, patients have usually transitioned out of the acute treatment phase and exhibit significant plasticity in physical and psychological recovery, making it a critical period for rehabilitation.
4. Severity of Stroke Sequelae: Stroke sequelae should be mild to moderate (Modified Rankin Scale score of 2 to 3). These patients have some level of independent mobility but still require rehabilitation training to further improve function.
5. Cognitive Ability: Participants must have basic cognitive function and be able to understand and comply with research requirements. This ensures that patients can effectively participate in art therapy and accurately report subjective experiences.
6. Emotional Status: Participants' levels of depression, anxiety, or stress should be mild to moderate at the start of the study. Patients with severe psychological disorders may require more intensive psychological support, which falls outside the scope of this study.
7. Language and Communication Skills: Participants must possess basic language expression and comprehension abilities to engage in and understand interactions during art therapy sessions. This ensures effective communication with the therapist.
8. Physical Condition: Participants must have the basic physical functions necessary to participate in art therapy, such as the ability to perform simple limb movements and activities. Severe physical disabilities may prevent participation in art activities.
9. Living Environment: Participants should reside in an area that allows them to regularly travel to the treatment site and have a relatively stable living environment. This helps ensure that patients can attend each therapy session on time and complete the entire intervention cycle.
10. Consent to Participate: Both the patient and their family members must fully understand the purpose, process, and potential risks of the study and be willing to sign an informed consent form. This ensures that patients fully comprehend their responsibilities and rights when participating in the study.
11. No Prior Psychological or Art Therapy: Participants must not have received any form of psychological therapy, art therapy, or similar rehabilitation intervention in the past 6 months to exclude the impact of other interventions on the study results.

Exclusion Criteria:

1. Severe Mental Illness: A history or current diagnosis of severe mental disorders (e.g., schizophrenia, bipolar disorder) or a current severe level of depression, anxiety, or stress. These mental health issues may require specialized psychological treatment, which is not aligned with the intervention objectives of this study.
2. Severe Comorbidities: Patients with serious physical illnesses, such as advanced cancer, severe heart disease (e.g., heart failure, acute coronary syndrome), chronic renal failure, or severe chronic respiratory diseases. These conditions may severely affect the patient's ability to participate and the rehabilitation outcomes.
3. Severe Sensory Impairments: Patients with serious sensory impairments, such as blindness, profound hearing loss, or uncorrectable sensory deficits. These impairments may prevent effective participation in art therapy, especially in activities requiring visual or auditory engagement (such as painting or music therapy).
4. Severe Language Impairments: Patients with severe aphasia or speech communication disorders that impede effective communication or expression. This would affect the patient's ability to participate in and understand the therapy process.
5. Substance Dependence or Abuse History: Patients with a current history of substance dependence or abuse (including alcohol and illicit drugs). Such conditions may significantly impact cognitive and behavioral functions, potentially interfering with the study's intervention effects.
6. Allergies or Physical Discomfort: Patients with severe allergic reactions to materials potentially used in art therapy (e.g., paint, clay, musical instruments) or a history of physical discomfort caused by similar materials.
7. Lack of Willingness to Participate: Patients or their family members show insufficient willingness to participate in the study or are unable to provide written informed consent. This may lead to premature withdrawal, affecting the study's integrity and result analysis.
8. Other Potential Influencing Factors: Any other factors not listed but considered by researchers to potentially affect patient participation or study outcomes. For example, significant life events (e.g., bereavement, divorce), which may have a considerable impact on the patient's psychological state.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Depression level | 1 month
  Hamilton Depression Rating Scale, 24-item version.The total score is 24 points, and the milder the disease, the lower the total score, the milder the degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuyuan People's Hospital, Jiamusi, Heilongjiang, China